CLINICAL TRIAL: NCT07335432
Title: Efficacy of Intravenous Vitamin C Versus Placebo on Estimated Blood Loss in Total Abdominal Hysterectomy
Brief Title: RCT - Efficacy of Intravenous Vitamin C Versus Placebo on Estimated Blood Loss in Total Abdominal Hysterectomy
Acronym: Vit C in TAH
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Principal Investigator, Aektanat Tawornkitpanich, M.D., Queen Savang Vadhana Memorial Hospital, Thailand
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 012/2567
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-09

CONDITIONS: Myoma;Uterus; Adenomyosis of Uterus
Keywords: Vitamin C; Total abdominal hysterectomy; Blood loss
MeSH Terms: conditions — Myofibroma; Adenomyosis; Hemorrhage | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Vitamin C (Experimental): Intervention Group: Received two 1 gm doses of Vitamin C intravenously (IV). first Dose: At midnight on the day of surgery. Second Dose: Immediately after the surgical incision. Control Group: Received two doses of a normal saline intravenously (IV) at the exact same times.
  Interventions: Dietary Supplement: Vitamin C (Ascorbic Acid)
- Placebo (Experimental)
  Interventions: Dietary Supplement: Vitamin C (Ascorbic Acid)

INTERVENTIONS:
Dietary Supplement: Vitamin C (Ascorbic Acid) — Received two 1 gm doses of Vitamin C intravenously (IV).
  first Dose: At midnight on the day of surgery.
  Second Dose: Immediately after the surgical incision.

SUMMARY:
Intervention Group: Received two 1 gm doses of Vitamin C intravenously (IV). first Dose: At midnight on the day of surgery. Second Dose: Immediately after the surgical incision. Control Group: Received two doses of a normal saline intravenously (IV) at the exact same times.

The primary outcome was to compare intraoperative blood loss between patients who received intravenous Vitamin C and those who did not, following an abdominal hysterectomy under general anesthesia.

Intraoperative estimated blood loss (EBL) was meticulously quantified by weighing surgical gauze and measuring suction canister volumes.

The secondary outcomes were to evaluate the potential benefits of Vitamin C administration, including:

* Reduction in the decline of hematocrit levels after surgery.
* Reduction of the length of hospital stay

ELIGIBILITY:
Inclusion Criteria:

* Female patients who underwent total abdominal hysterectomy

  * No bleeding tendency.
  * No history of anticoagulant or thrombolytic drug use
  * No contraindications to vitamin C supplementation

Exclusion Criteria:

* Inability to communicate in the Thai language.

  * Underwent total abdominal hysterectomy due to gynecologic malignancy.
  * Required emergency total abdominal hysterectomy.
  * History of vitamin C supplementation within 2 weeks prior to surgery.
  * History of smoking.
  * Previous abdominal surgery, such as bowel surgery, cesarean section

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative estimate blood loss | intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Savang Vadhana Memorial hospital, Si Racha, Changwat Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Data was save in form of microsoft excel spreadsheet and SPSS file